CLINICAL TRIAL: NCT04945226
Title: A Randomized, Open-Label, Exploratory, Pharmacokinetic, Sequential Single Ascending Dose Study of IVL3001 Versus Propecia (Finasteride) Tablets in Healthy Adult Participants
Brief Title: A Clinical Trial to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of IVL3001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inventage Lab., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IVL3001-001
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Finasteride; Tablets

STUDY DESIGN:
Intervention Model Description: Cohort 1 / Cohort 2 (Group 1, Group 2) / Cohort 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propecia (Active Comparator): Propecia Tablet, QD, PO
  Interventions: Drug: Finasteride 1mg Tablet
- IVL3001 (A mg) (Experimental): S.C, Single Dose.
  Interventions: Drug: IVL3001
- IVL3001 (B mg) (Experimental): S.C, Single Dose.
  Interventions: Drug: IVL3001
- IVL3001 (C mg) (Experimental): S.C, Single Dose.
  Interventions: Drug: IVL3001

INTERVENTIONS:
Drug: Finasteride 1mg Tablet — Propecia Tablet 1mg
  Arms: Propecia
Drug: IVL3001 — Finasteride long acting injection
  Arms: IVL3001 (A mg); IVL3001 (B mg); IVL3001 (C mg)

SUMMARY:
A Clinical Trial to Assess Pharmacokinetic/Pharmacodynamic Profiles and Safety of IVL3001

DETAILED DESCRIPTION:
A Randomized, Open-Label, Exploratory, Pharmacokinetic, Sequential Single Ascending dose Study of IVL3001 Versus Propecia (Finasteride) Tablets in Healthy Adult Participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, non-smoker or, if a moderate or occasional smoker (< 10 cigarettes per day or nicotine equivalent) must agree to abstain from smoking from 48 h before first IP administration through to completion of the final EOS/ET visit, aged ≥ 18 to 55 years (inclusive at the time of informed consent)
* In good general health, in the opinion of the Investigator, with no significant medical history, and have no clinically significant abnormalities on complete physical examination, 12-lead ECG, heart rate, and BP, both at Screening and before administration of the initial dose of IP
* Body mass index (BMI) between ≥ 18 kg/m2 and ≤ 32 kg/m2 and a minimum weight ≥ 50 kg and ≤ 100 kg at Screening
* Clinical laboratory values within normal limits, with normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate
* Ability and willingness to attend the necessary visits to the CRU and be domiciled overnight
* Willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any protocol-specific study procedures

Exclusion Criteria:

* Prior or ongoing medical conditions, medical history, physical examination findings, or laboratory abnormalities that, in the Investigator's (or delegate's) opinion, could adversely affect the safety of the participant
* Presence or history of any clinically significant blood, kidney, endocrine, lung, gastrointestinal tract, cardiovascular, liver, or neurological condition
* Presence of any underlying physical or psychological (eg, depression) medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol. Mild depression and anxiety that has been resolved at least 6-12 months ago is accepted.
* Presence of any medical condition that may affect oral drug absorption (eg, gastrectomy, gall bladder removal, bariatric surgery, gastric bypass and sleeve, bowel resection)
* Hypersensitivity to finasteride or to any excipient of the IPs
* Age adjusted PSA between 0 2.5 ng/mL for subjects ≤ 50 years of age and between 0-4 ng/mL for subjects > 50 years of age at Screening, unless deemed not clinically significant by the Investigator or delegate
* History or known presence of any prostatic problem (infection, prostate cancer, stricture disease, hypotonic bladder or other neurogenic disorder that might mimic BPH)
* Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), HIV antigen or antibody at Screening
* Positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, benzodiazepines, opiates and cocaine), or a positive alcohol breath (or urine), or cotinine test
* History of alcohol or substance abuse or dependency, or history of recreational intravenous (IV) drug use over the last 1 year (by self-declaration)
* Regular alcohol consumption defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit, or a 125 mL glass of wine) within 6 months of Screening.
* Use of any IP or investigational medical device within 3 months prior to Screening, or five half-lives of the product (whichever is the longest), or participation in more than 4 investigational drug studies within 1 year prior to Screening
* Use of any drug known to significantly induce or inhibit drug absorption or metabolism within 30 days prior to dosing
* An employee, or relative of an employee, directly involved in the conduct of the study
* Unwilling to refrain from strenuous exercise from 48 hours prior to admission to the CRU at Day -1 and 48 hours prior to each follow-up
* Presence of sexual dysfunction such as decreased libido, erectile dysfunction, or ejaculation disorder
* Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2 at Screening
* Any reason which, in the opinion of the PI, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
AUClast of IVL3001 | Pre-dose, 1008 hours
  Area under the concentration-time curve from time zero to last
AUCinf of IVL3001 | Pre-dose, 1008 hours
  Area under the concentration-time curve from time zero to infinity
AUC0-1008h of IVL3001 | Pre-dose, 1008 hours
  Area under the concentration-time curve from time zero to 1008 hours
AUClast of Propecia | Pre-dose, 816 hours
  Area under the concentration-time curve from time zero to last
AUCinf of Propecia | Pre-dose, 816 hours
  Area under the concentration-time curve from time zero to infinity
AUC0-672h of Propecia | Pre-dose, 672 hours
  Area under the concentration-time curve from time zero to 672hours

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Brisbane, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Ryu C, Lee M, Lee KR, Kim J. A Phase I, Open-Label, Sequential, Single-Dose Clinical Trial to Evaluate the Pharmacokinetic, Pharmacodynamic, and Safety of IVL3001, a Finasteride-Based Novel Long-Acting Injection for Androgenetic Alopecia. Adv Ther. 2024 Jul;41(7):2936-2952. doi: 10.1007/s12325-024-02890-1. Epub 2024 Jun 4. PMID 38833144